CLINICAL TRIAL: NCT06060210
Title: Impact of Ketamine On Depressive Symptoms In Patients Undergoing Lumbo-peritoneal Shunt Insertion. A Randomized Double-blind Controlled Trial.
Brief Title: Impact of Ketamine On Depressive Symptoms In Patients Undergoing Lumbo-peritoneal Shunt Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Abdel Fatah, lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC 12-9-2023
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2024-12

CONDITIONS: Depression, Anxiety
Keywords: ketamine; perioperative depression; lumboperitoneal shunt
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Saline Solution; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): 50-ml volume of normal saline
  Interventions: Drug: normal Saline
- Group B (Active Comparator): 50-ml volumes, and the ketamine concentration is 1 mg/ml
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: normal Saline — 50-ml Saline
  Arms: Group A
Drug: Ketamine — 50-ml volumes, and the ketamine concentration is 1 mg/ml
  Other Names: katalar
  Arms: Group B

SUMMARY:
Postoperative depression is a perioperative psychological complication that severely affects patient recovery and quality of life. In extreme cases, it may lead to suicidal behavior. Postoperative depression can be seen in various surgical operations .

High rates of anxiety and depression have been reported in cohorts of patients with IIH, though it is not clear whether there is any direct relationship. Worse outcomes in terms of disability level and symptom resolution have been observed in IIH patients who have a known co-existing psychiatric illness compared to those who do not .

DETAILED DESCRIPTION:
Postoperative depression is a perioperative psychological complication that severely affects patient recovery and quality of life. In extreme cases, it may lead to suicidal behavior. Postoperative depression can be seen in various surgical operations.

Idiopathic intracranial hypertension (IIH) is the most common cause of papilledema and is typically seen in young women with elevated body mass index. The prevalence of IIH has been increasing in recent years, in parallel with climbing rates of obesity .

High rates of anxiety and depression have been reported in cohorts of patients with IIH, though it is not clear whether there is any direct relationship. Worse outcomes in terms of disability level and symptom resolution have been observed in IIH patients who have a known co-existing psychiatric illness compared to those who do not .

The use of lumbo-peritoneal (LP) shunts has been well documented as a treatment modality for patients with idiopathic intracranial hypertension (IIH). There are a number of advantages to LP shunts when compared with other treatment modalities for IIH, such as stereotactic ventriculo-peritoneal shunts (VP) and optic nerve sheath fenestrations (ONSF). LP shunts avoid intracranial risks, such as cerebral hemorrhage, seizures, and shunt malposition.

Over the past decade, it has been provoked a single administration of ketamine elicits fast (in as little as half an hour) and sustained antidepressant effects both in human and animal models of depression. There are some potential mechanisms of antidepressant actions of ketamine. MK-801, a noncompetitive NMDA receptor antagonist, produced antidepressant-like actions in the animal model of depression . Ketamine can also increase hippocampal brain-derived neurotrophic factor levels, which may be important for producing a rapid onset of antidepressant action .A recent study found ketamine could quickly elevate mood by blocking NMDAR receptor-dependent bursting activity of the lateral habenula neurons to disinhibit downstream monoaminergic reward centers and provide a framework for developing new rapid-acting antidepressants .

Accordingly, we hypothesized that intraoperative ketamine can reduce the post operative depressive symptoms after theco-peritoneal shunt insertion.

ELIGIBILITY:
Inclusion Criteria:

* patients of both sex
* with an age range from 20 to 44 years old
* having moderate to severe depressive symptoms
* an expected hospital stay of no less than 7 days

Exclusion Criteria:

* history of epilepsy
* major depressive disorder patients
* drug abuse
* history of allergy to the research drug
* heart rate > 120 beats per minute
* systolic blood pressure > 180 mmHg
* heart failure
* renal or liver dysfunction
* patients who cannot cooperate to complete psychiatric assessments
* pregnant or breast-feeding women
* patients who refuse to sign informed consent.

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2023-10-29 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
the rate of response to treating postoperative depression | at 3 postoperative days
  defined as a relative reduction of more than 50% from the baseline 10-item MADRS score

SECONDARY OUTCOMES:
The remission rate | at 1 and 3 days after the administration of ketamine.
  defined as an absolute value of MADRS score of no more than 10
The incidence of severe pain | within the first 48 hours postoperatively
  From 0 to 10 (0 no pain , 10 very sever pain)
The quality of life | within 7 days postoperatively
  a scale ranging from 100-0, where 100 is labeled 'Perfect quality of life,' and 0 is labeled 'Might as well be dead'.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ah Abdelfatah, MD, Principal Investigator — banha faculity of medicine
Locations (1):
- Banha faculity of medicine, Banhā, Elqalyoubea, Egypt